CLINICAL TRIAL: NCT06272409
Title: Phase III, Multicenter, Double-blind, Planned, Parallel Clinical Trial to Evaluate the Efficacy and Safety of DEP114 in the Treatment of Moderate to Severe Persistent Allergic Rhinitis in Children Aged Between 6 and 11 Years
Brief Title: Efficacy and Safety of DEP114 in the Treatment of Moderate to Severe Persistent Allergic Rhinitis in Children.
Acronym: SIERRA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEP114-III-0123
Record Dates: First submitted 2024-02-09; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEP114 (Experimental): DEP114 administered once (01) time a day, by morning, for 5 (+2) days.
  Interventions: Drug: DEP114
- DESLORATADINE (Active Comparator): Desloratadine administered once (01) time a day, by morning, for 5 (+2) days.
  Interventions: Drug: Desloratadine 0.5 MG/ML

INTERVENTIONS:
Drug: DEP114 — DEP114 oral solution
  Arms: DEP114
Drug: Desloratadine 0.5 MG/ML — Desloratadine oral solution
  Arms: DESLORATADINE

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of DEP114 in the treatment of Moderate to Severe Persistent Allergic Rhinitis in children aged between 6 and 11 years.

DETAILED DESCRIPTION:
* double-blind, superiority, parallel group trial.
* Experiment duration: 05 days.
* 03 visits (days 0, 5 and 28).
* Efficacy will be evaluated for persistent allergic rhinitis based on Global improvement in nasal symptoms score
* Adverse events evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree for all the purposes of the test, signing and dating the Term of Free and Informed Assent (TALE), signed by the Free and Informed Consent Form (TCLE) by responsible;
* Age ≥ 6 years and ≤ 11 years on the day of signing the TALE and the TCLE by the person responsible;
* Diagnosis of moderate to severe persistent allergic rhinitis (PAR) according to the criteria of Allergic Rhinitis and its Impact on Asthma (ARIA);
* Presence of sensitization to aeroallergens confirmed by positive result to the immediate reading skin test (PRICK test) and/or the presence of specific IgE to the test radioallergoabsorbent (RAST);
* Symptom intensity score "nasal obstruction" ≥ 2 points.
* Total nasal symptoms score (TNSS) ≥ 8 points.

Exclusion Criteria:

* Use of prednisolone or other oral or parenteral corticosteroid in the seven (07) days prior to inclusion;
* Use of H1 antihistamine, anti-leukotriene and decongestant topic in the seven (07) days prior to inclusion;
* Use or indication for the use of antibiotics at the screening visit and randomization;
* Presence of adenoid hypertrophy or anatomical disorders known obstructive disorders (e.g. septal deviation) that may be held responsible for nasal obstruction, at the discretion of the investigator;
* Diagnosis of severe or uncontrolled asthma;
* Allergy to desloratadine, prednisolone or any other component of the formulation of investigational products (PSIs);
* Presence of systemic fungal infection;
* Presence of any uncontrolled infection;
* Presence of any clinical observation finding (evaluation clinical/physical) or laboratory condition that is interpreted by the investigator physician as a risk to participation in the trial clinical or presence of serious uncontrolled disease(s);
* Participants who are pregnant or breastfeeding;
* Participation in clinical trial protocols in the last 12 (twelve) months (CNS Resolution 251, of August 7, 1997, item III, subitem J), unless the investigator believes that there may be direct benefit to the participant.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the superiority of DEP114 in relation to desloratadine 0.5 mg/mL in relieving the nasal symptoms of moderate to severe persistent allergic rhinitis in children, five days after starting treatment. | 5 days
  Global improvement in nasal symptoms (absolute variation in total nasal symptoms score obstruction, runny nose, itching and sneezing, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms and 3=severe symptoms) five days after the start of treatment.

SECONDARY OUTCOMES:
To evaluate the effectiveness of DEP114 in relieving nasal symptoms of moderate to severe persistent allergic rhinitis in children, throughout the treatment. | 1-5 days
  Global improvement in nasal symptoms throughout treatment (absolute variation in the total score of nasal symptoms, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms and 3=severe symptoms) on days 1, 2, 3, 4 and 5.
  Improvement of nasal symptoms three days after the start of the treatment (proportion of participants with improvement in total nasal symptoms score, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms and 3=severe symptoms) three days after the start of treatment, with improvement in total nasal symptoms score change of at least 4 points on day 3 compared to at baseline).
Evaluate the efficacy of DEP114 to relieve nasal obstruction present in moderate to severe persistent allergic rhinitis in children through the treatment. | 1-5 days
  Improvement of nasal obstruction throughout treatment (absolute variation in total nasal symptoms score obstruction, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms and 3=severe symptoms) on days 1, 2, 3, 4 and 5.
Evaluate the efficacy of DEP114 to relieve coryza present in moderate to severe persistent allergic rhinitis in children, three and five days after the start of treatment. | 3 and 5 day
  Improvement of the runny nose three and five days after the start of the treatment (distribution of participants according to intensity of coryza at baseline, three and five days after the start of treatment).
Evaluate the efficacy of DEP114 to relieve nasal itching present in moderate to severe persistent allergic rhinitis in children, three and five days after the start of treatment. | 3 and 5 day
  Improvement of nasal itching three and five days after the onset treatment (distribution of participants according to intensity of nasal itching at baseline, three and five days after starting treatment).
Evaluate the efficacy of DEP114 to relieve sneezing present in persistent allergic rhinitis moderate to severe in children, three and five days after the start of treatment. | 3 and 5 day
  Improvement in sneezing three and five days after the start of the treatment (distribution of participants according to intensity of sneezing at baseline, three and five days after starting treatment).
Evaluate the efficacy of DEP114 to relieve symptoms of moderate to severe persistent allergic rhinitis in children according to the perception of the person responsible for the participant. | 5 day
  Overall assessment of the treatment by the person responsible for the treatment participant five days after the start of treatment (distribution of participants according to a 5-point categorical scale, where 0=very bad, 1=bad, 2=neither good nor bad, 3=good, 4=very good).
Evaluate the efficacy of DEP114 to relieve symptoms of moderate to severe persistent allergic rhinitis in children according to the investigator's perception. | 5 day
  Overall assessment of treatment by the investigator five days after the start of treatment (distribution of participants according to a 5-point categorical scale, where 0=very bad 1=bad, 2=neither good nor bad, 3=good, 4=very good).